CLINICAL TRIAL: NCT00378664
Title: Lumbar to Sacral Ventral Nerve Re-Routing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-124
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Urinary Incontinence; Spinal Cord Injury; Spina Bifida
Keywords: urinary incontinence; spinal cord injury; spina bifida
MeSH Terms: conditions — Urinary Incontinence; Spinal Cord Injuries; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): All enrollees are included in the intervention - lumbar to sacral ventral nerve re-routing procedure surgical nerve re-routing procedure.
  Interventions: Procedure: lumbar to sacral ventral nerve re-routing procedure

INTERVENTIONS:
Procedure: lumbar to sacral ventral nerve re-routing procedure — surgical nerve re-routing procedure

SUMMARY:
To assess the level of improvement in voiding function after lumbar to sacral ventral nerve re-routing procedure in Spinal Cord Injury and spina bifida patients

DETAILED DESCRIPTION:
Spinal cord injury (SCI) and spina bifida is a source of irreversible injury to the spinal cord often resulting in paralysis and loss of sensation below the waist. The inability to urinate normally is a consequence of both conditions (neurogenic voiding dysfunction). In spina bifida and spinal cord injury, the nerve that controls the bladder and sphincter (the muscle that squeezes the bladder neck to prevent leaking) may no longer work properly resulting in patients who cannot urinate or are constantly wet.

Most patients will maintain high pressures in their bladder and these elevated pressures will eventually take its toll by causing recurrent urinary tract infections, backup of urine to the kidneys, and marked dilatation of possible further damage to the kidneys. Many patients eventually suffer from irreversible renal (kidney) damage, where dialysis or kidney transplant is the only way to sustain life.

Spinal bifida (present at birth) and SCI (occurs most often early in the fourth decade of life) predominately affect young individuals and longevity and quality of life may be greatly reduced by the presence of bladder, bowel, and sexual dysfunction. In the recent past, medications and catheters were the only way to help cord injured patients empty their bladders. Although clean intermittent catheterization (CIC) provides good maintenance results, medications can help conserve low bladder pressures, and antibiotics sustain an infection free urinary tract, these are difficult bladder management programs to uphold. They are expensive, time consuming, and outcomes are inconsistent.

A new surgical procedure has potential for treatment of spinal cord injuries/ spinal bifida. Recently, Dr. Chuan-Guo Xiao from China developed a surgical procedure of rewiring the nerves in the spinal cord to gain better control of urination and avoid complications of neurogenic bladder. The procedure reconnects live wires (nerves) to dead wires.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female paraplegics 18 years and older with spinal cord lesion above L1 on a CIC program for bladder management and a score of "A" on ASIA scale.
2. Male and female patients age 6 and older with myelomeningocele spina bifida (surgically closed at birth) on a CIC program for bladder management.
3. Neurogenic bladder documented by urodynamic testing.
4. Stable neurogenic bladder dysfunction of at least 1 year or more.
5. Compliant bladder wall.
6. Normal renal function.

Exclusion Criteria:

1. History of bladder cancer, augmentation, or radiation.
2. Bladder capacity less than 100 milliliters (ml).
3. Anatomic outlet obstruction or urethral strictures.
4. Vesico-ureteric reflux grade 2 or higher.
5. Presence of an ileal conduit or supra-pubic catheter drainage.
6. Contraindications to general anesthesia or surgery.
7. Inability to complete follow up visits for 3 years.
8. Inability to comprehend and answer self-administered questionnaires.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assess the level of improvement in voiding function after lumbar to sacral ventral nerve re-routing procedure in SCI and spina bifida patients. | evaluated at 6 months and 1 year

SECONDARY OUTCOMES:
Assess the effect of lumbar to sacral ventral the nerve re-routing on bowel function in SCI and spina bifida patients | evaluated at 6 month and 1 year visit
Assess the effect of the lumbar to sacral ventral nerve re-routing on health related quality of life in SCI and spina bifida patients | evaluate at 6 month and 1 year
Assess the effect of the lumbar to sacral ventral nerve re-routing on ability to perform activities of daily living in SCI and spina bifida patients | evaluate at 6 month and 1 year visit
Assess the effect of the lumbar to sacral ventral nerve re-routing on sexual function in SCI patients 18 years of age and older | evaluate at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, M.D., Principal Investigator — Corewell Health East

REFERENCES:
- [Background] Xiao CG. Reinnervation for neurogenic bladder: historic review and introduction of a somatic-autonomic reflex pathway procedure for patients with spinal cord injury or spina bifida. Eur Urol. 2006 Jan;49(1):22-8; discussion 28-9. doi: 10.1016/j.eururo.2005.10.004. Epub 2005 Nov 2. PMID 16314037
- [Background] Liu Z, Liu CJ, Hu XW, Du MX, Xiao CG. [An electrophysiological study on the artificial somato-autonomic pathway for inducing voiding]. Zhonghua Yi Xue Za Zhi. 2005 May 25;85(19):1315-8. Chinese. PMID 16029629
- [Background] Mathews TJ, Honein MA, Erickson JD. Spina bifida and anencephaly prevalence--United States, 1991-2001. MMWR Recomm Rep. 2002 Sep 13;51(RR-13):9-11. PMID 12353510
- [Background] Muller T, Arbeiter K, Aufricht C. Renal function in meningomyelocele: risk factors, chronic renal failure, renal replacement therapy and transplantation. Curr Opin Urol. 2002 Nov;12(6):479-84. doi: 10.1097/00042307-200211000-00006. PMID 12409876
- [Derived] Peters KM, Gilmer H, Feber K, Girdler BJ, Nantau W, Trock G, Killinger KA, Boura JA. US Pilot Study of Lumbar to Sacral Nerve Rerouting to Restore Voiding and Bowel Function in Spina Bifida: 3-Year Experience. Adv Urol. 2014;2014:863209. doi: 10.1155/2014/863209. Epub 2014 Jun 2. PMID 24987412